CLINICAL TRIAL: NCT04875975
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase 2 Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Rozanolixizumab in Adult Study Participants With Leucine-Rich Glioma Inactivated 1 Autoimmune Encephalitis
Brief Title: A Study to Test the Efficacy, Safety, and Pharmacokinetics of Rozanolixizumab in Adult Study Participants With Leucine-Rich Glioma Inactivated 1 Autoimmune Encephalitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study stopped prematurely due to enrolment challenges, the termination was not linked to any safety issues.
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AIE001; 2019-004778-25 (EudraCT Number)
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Leucine-Rich Glioma Inactivated 1 Autoimmune Encephalitis
Keywords: Leucine-Rich Glioma Inactivated 1 Autoimmune Encephalitis; Phase 2; Rozanolixizumab
MeSH Terms: interventions — rozanolixizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rozanolixizumab (Experimental): Participants will be randomized to receive a predefined dose of rozanolixizumab.
  Interventions: Drug: Rozanolixizumab
- Placebo (Placebo Comparator): Participants will be randomized to receive a dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rozanolixizumab — * Pharmaceutical form: Solution for infusion
  * Route of administration: Subcutaneous use
  Subjects will receive rozanolixizumab in a pre-specified sequence during the Treatment Period.
  Arms: Rozanolixizumab
Drug: Placebo — * Pharmaceutical form: Solution for infusion
  * Route of administration: Subcutaneous use
  Subjects will receive placebo in a pre-specified sequence during the Treatment Period.
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the efficacy of rozanolixizumab as measured by seizure freedom, change in cognitive function, use of rescue medication, onset of seizure freedom and to assess safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be ≥18 to ≤89 years of age
* Study participant must be seropositive for leucine-rich glioma inactivated 1 (LGI1) antibody
* Study participant must have ≥2 seizures/week during the Screening Period or have experienced such seizures that stopped following high dose corticosteroids (500 to 1000 milligram (mg) methylprednisolone (MP) equivalent/day):

  * Either faciobrachial dystonic seizures (FBDS) with or without other focal (partial) seizures including focal to bilateral tonic clonic
  * Or focal (partial) seizures including focal to bilateral tonic clonic and fulfil the following new-onset Autoimmune encephalitis (AIE) criteria
* Study participant has initiated or re-initiated corticosteroids at a dose of 500 to 1000 mg MP equivalent/day within 42 days prior to randomization. Participants re-initiating corticosteroids are eligible only if re-initiation is due to seizure rebound and within the timeframe outlined. If the study participant has initiated a steroid taper, the study participant cannot receive an oral steroid dose lower than 40mg/day when randomized
* Study participant with onset of disease symptom between 0 to 12 months prior to Screening, per investigator's assessment.
* Study participant weighs at least 35 kg at Screening
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  i) Not a woman of childbearing potential (WOCBP) OR ii) A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 90 days after the final dose of study treatment

Exclusion Criteria:

* Study participant has a known hypersensitivity to any components of the study medication or any other anti-neonatal Fc receptor (FcRn) medications.
* Study participant has a confirmed prior diagnosis of epilepsy or new onset seizures that are unrelated to LGI1 autoimmune encephalitis (AIE) or has any known or suspected medical cause for the onset of seizures other than possible AIE
* Study participant has a known active neoplastic disease or history of neoplastic disease within 5 years of study entry
* Study participant has renal impairment, defined as glomerular filtration rate (GFR) <30mL/min/1.73m2 at the Screening Visit
* Study participant has a clinically important active infection (including unresolved or not adequately treated infection) as assessed by investigator, including participants with a serious infection within 6 weeks prior to the first dose of investigational medicinal product (IMP)
* Study participant has a history of chronic ongoing infections
* Study participant has current unstable liver or biliary disease, per investigator assessment, defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis
* Study participant has positive tuberculosis (TB) test at the Screening Visit
* Study participant has a history of solid organ transplant or hematopoietic stem cell transplant
* Study participant has undergone a splenectomy
* Study participant has a current or medical history of primary immune deficiency
* Study participant has received a live vaccination within 4 weeks prior to the Baseline Visit; or intends to have a live vaccination during the course of the study or within 8 weeks following the final dose of investigational medicinal product (IMP)
* Study participant has previously received rozanolixizumab drug product
* Alanine transaminase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) are >3x upper limit of normal (ULN)
* Study participant has a total IgG level ≤5.5 g/L at the Screening Visit
* Study participant has absolute neutrophil count <1500 cells/mm^3 at the Screening Visit

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (27):
- United States (9):
  - Aie001 50101, Aurora, Colorado
  - Aie001 50342, Jacksonville, Florida
  - Aie001 50243, Boston, Massachusetts
  - Aie001 50047, Boston, Massachusetts
  - Aie001 50104, Rochester, Minnesota
  - Aie001 50298, New York, New York
  - Aie001 50090, Winston-Salem, North Carolina
  - Aie001 50311, Cleveland, Ohio
  - Aie001 50304, Dallas, Texas
- Aie001 30027, Melbourne, Australia
- Aie001 40123, Brussels, Belgium
- France (7):
  - Aie001 40129, Bordeaux
  - Aie001 40426, Bron
  - Aie001 40364, Lille
  - Aie001 40546, Nancy
  - Aie001 40132, Nice
  - Aie001 40019, Paris
  - Aie001 40286, Toulouse
- Germany (2):
  - Aie001 40515, Berlin
  - Aie001 40249, Kiel
- Italy (2):
  - Aie001 40695, Pavia
  - Aie001 40567, Roma
- Aie001 40264, Rotterdam, Netherlands
- Spain (2):
  - Aie001 40267, Barcelona
  - Aie001 40341, Málaga
- United Kingdom (2):
  - Aie001 40168, Nottingham
  - Aie001 40163, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in September 2021 and concluded in April 2024.
Pre-assignment Details: The Participant Flow refers to the Randomized Set (RS).
Groups:
- Placebo: Participants received placebo as a subcutaneous (sc) infusion once a week (Q1W) for 25 weeks.
- Rozanolixizumab (RLZ): Participants received rozanolixizumab as a sc infusion Q1W for 25 weeks.
Period: Overall Study
Arm/Group | Placebo | Rozanolixizumab (RLZ)
Started | 6 | 6
Completed | 2 | 0
Not Completed | 4 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 2 | 2
Not completed — Permanently left due to seizure recurrence | 1 | 0
Not completed — Relapse With Insults | 0 | 1
Not completed — Permanently left due to new seizure recurrence | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set (RS) which consisted of all enrolled study participants who were randomized to treatment arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rozanolixizumab (RLZ) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (12.4) | 70.7 (11.4) | 65.7 (12.5)
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 years | 3 | 1 | 4
  65 - <85 years | 3 | 5 | 8
  >=85 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 4 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 4 | 9
  Missing | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 5 | 4 | 9
  Missing | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Seizure Free Study Participants at the End of the Treatment
Description: Seizure freedom was defined as a minimum of 28 consecutive days of no seizures of any type during the treatment and maintained until the end of the treatment (Week 25).
Time Frame: From Baseline until the end of the Treatment (Week 25)
Population: The Randomized Set (RS) consisted of all enrolled study participants who were randomized to treatment arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rozanolixizumab (RLZ)
Number analyzed (Participants) | 6 | 6
Participants | 1 | 0

2. Secondary Outcome: Change From Baseline in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Total Scale Index Score at the End of the Treatment
Description: The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) consists of 12 subtests that contribute to 5 age-based domain index scores (immediate memory, visuospatial/constructional, language, attention, delayed memory) that were aggregated for a total scale index score. All index scores have an age-based mean of 100, with a standard deviation (SD) of 15. The total scale score was calculated by taking the mean of the sum of the five index scores. Total possible scale index scores range from 40-135. Higher scores reflect better neurocognitive performance. The total scale index score is the score typically used to reflect global neurocognitive status. Baseline of RBANS is defined as the screening (Visit 1, Week -1) value.
Time Frame: From Baseline to Week 5, 13, 21 and 25
Population: The Randomized Set (RS) consisted of all enrolled study participants who were randomized to treatment arms. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure. Here, number analyzed signifies participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rozanolixizumab (RLZ)
Number analyzed (Participants) | 4 | 6
score on a scale
  Week 5 | 4.5 (2.6) | 2.2 (11.3)
  Week 13: number analyzed (Participants) | 4 | 4
  Week 13 | 7.0 (2.9) | 12.3 (7.9)
  Week 21: number analyzed (Participants) | 4 | 2
  Week 21 | 7.0 (7.3) | NA (NA) — As pre-specified in the SAP, mean and SD will only be calculated if number of participants are equal to 3 or greater than 3. Here, Mean and SD were not calculated due to less than 3 participants.
  Week 25: number analyzed (Participants) | 2 | 1
  Week 25 | NA (NA) — As pre-specified in the SAP, mean and SD will only be calculated if number of participants are equal to 3 or greater than 3. Here, Mean and SD were not calculated due to less than 3 participants. | NA (NA) — As pre-specified in the SAP, mean and SD will only be calculated if number of participants are equal to 3 or greater than 3. Here, Mean and SD were not calculated due to less than 3 participants.

3. Secondary Outcome: Percentage of Participants With a Favorable Outcome in the Modified Rankin Scale (mRS) During the Treatment
Description: Percentage of participants with a favorable outcome in mRS during treatment, where favorable outcome defined as no worsening for participants with Baseline mRS score of ≤1 or improvement of ≥1 point for participants with Baseline mRS score of ≥2. The mRS is commonly used scale for measuring degree of disability or dependence in daily activities of people who suffered a stroke or other causes of neurological disability. The scale ranges from 0 (perfect health) to 6 (death).
  0-No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk and attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Time Frame: From Baseline until the end of the Treatment (Week 25)
Population: The Randomized Set (RS) consisted of all enrolled study participants who were randomized to treatment arms. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure. Analysis datasets were not generated an output when the n < 3, therefore, no data obtained and reported.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rozanolixizumab (RLZ)
Number analyzed (Participants) | 2 | 1
percentage of participants | NA — Analysis datasets were not generated an output when the n < 3, therefore, no data obtained and reported. | NA — Analysis datasets were not generated an output when the n < 3, therefore, no data obtained and reported.

4. Secondary Outcome: Number of Participants Who Required Rescue Medication Due to an Absence or Loss of Clinical Benefit During the Treatment
Description: Study participants who required rescue medication due to an absence or loss of clinical benefit were discontinued blinded treatment and completed the assessments for the early discontinuation visit.
Time Frame: From Baseline until the end of the Treatment (Week 25)
Population: The Randomized Set (RS) consisted of all enrolled study participants who were randomized to treatment arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rozanolixizumab (RLZ)
Number analyzed (Participants) | 6 | 6
Participants | 3 | 2

5. Secondary Outcome: Time to First Occurrence of Seizure Freedom During the Treatment
Description: The time to first occurrence of seizure freedom was defined by the number of days after randomization to the first day of the first 28 consecutive days without seizures during the treatment. Time to first occurrence of 28 consecutive days of seizure freedom (days) during the treatment was calculated as date of first day of occurrence of 28 consecutive days of seizure freedom - Date of Randomization + 1.
Time Frame: From Baseline until the end of the Treatment (Week 25)
Population: The Randomized Set (RS) consisted of all enrolled study participants who were randomized to treatment arms.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Placebo | Rozanolixizumab (RLZ)
Number analyzed (Participants) | 6 | 6
Weeks | 0.1 [0.1 to 8.4] | 0.1 [0.1 to 8.3]

6. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP, whether or not related to the IMP. A TEAE was defined as an AE starting on or after the time of first administration of IMP or any unresolved event already present before the first administration of IMP that worsens in intensity following exposure to treatment up to the end of the Treatment and including the 8-week (56 days) Safety-Follow Up (SFU).
Time Frame: From Baseline until the End of Study (Week 32)
Population: The Safety Set (SS) consisted of all randomized study participants who received at least one dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rozanolixizumab (RLZ)
Number analyzed (Participants) | 6 | 6
percentage of participants | 100 | 100

ADVERSE EVENTS:
Time Frame: From Baseline until the End of Study (up to Week 32)
Description: A TEAE was defined as an AE starting on or after the time of first administration of IMP or any unresolved event already present before the first administration of IMP that worsens in intensity following exposure to treatment up to the end of the Treatment and including the 8-week (56 days) SFU. The Safety Set consisted of all randomized study participants who received at least one dose of IMP.
Arm/Group | Placebo | Rozanolixizumab (RLZ)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Rozanolixizumab (RLZ) (N=6)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Psoas abscess (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Rozanolixizumab (RLZ) (N=6)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 3 (7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 2 (2) | 0 (0)
Swelling face (General disorders) | 0 (0) | 1 (1)
Infusion site erythema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 4 (4)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood immunoglobulin M increased (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (4) | 1 (1)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Affect lability (Psychiatric disorders) | 0 (0) | 1 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (3)
Emotional disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Impulse-control disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (2)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the early termination of the recruitment and insufficient participants, it was not feasible to carry out the statistical analyses as originally planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT04875975/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT04875975/SAP_001.pdf